CLINICAL TRIAL: NCT06831032
Title: A Phase I, Prospective, Single-Arm Feasibility Study: Elective Adaptive Radiation With SBRT for Improved DurabilitY of Response (EASY)
Brief Title: Elective Adaptive Radiation With SBRT for Improved DurabilitY of Response
Acronym: EASY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-6066
Record Dates: First submitted 2025-02-13; First posted 2025-02-17 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Prostate Adenocarcinoma; Iliac Nodal Disease; Para-aortic Lymph Node Metastasis; Para-aortic Nodal Disease; Oligorecurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT delivered with CBCT-guided online adaptive RT (Experimental): Patients will undergo CT guided online adaptive SBRT 30-40Gy to the tumor nodal GTV volume(s) plus 25Gy in 5 fractions ENI to PA nodes (+/- pelvic nodes).
  Interventions: Radiation: Adaptive radiotherapy using SBRT

INTERVENTIONS:
Radiation: Adaptive radiotherapy using SBRT — Adaptive External beam radiotherapy using SBRT 30-40Gy to the tumor nodal GTV volume(s) plus 25 Gy in 5 fractions ENI to PA nodes (+ common iliac nodes)

SUMMARY:
This prospective, single-arm feasibility study will include patients with prostate cancer that have controlled local disease diagnosed with oligorecurrent para-aortic nodal disease and/or common iliac nodal disease detected by PSMA PET or conventional CT/MRI imaging, and these patients will undergo CT-guided online adaptive SBRT to the tumor and elective SBRT to adjacent at-risk nodal regions.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed prostate adenocarcinoma.
2. Oligorecurrent para-aortic +/- common iliac nodal disease planned for SBRT.
3. ≤10 involved para-aortic (defined as between L1/L2 interface and L4/L5 interface) +/- common iliac LN on PSMA PET imaging.
4. ECOG performance status 0-2.

Exclusion Criteria:

1. Prior radiotherapy to the nodal echelon (PA +/- common iliac).
2. Active secondary malignancy, except for adequately treated non-melanoma skin cancer.
3. Presence of significant comorbidities or medical conditions that may compromise the ability to undergo radiotherapy or participate in the study.
4. Contraindication to radiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Quantify adverse events using CTCAE v5.0 | 2 years
  Acute toxicities (≤3 months) and long-term toxicities (related to urinary, bowel or sexual function) will be collected and evaluated by the CTCAE v5.0.

SECONDARY OUTCOMES:
QoL using EPIC questionnaire | 2 years
  Quality of life (QOL) will be collected using expanded prostate cancer index composite (EPIC) questionnaire. The quality-of-life scores will be converted to a scale of 0-100 for each category. A higher score indicates a better quality of life.
Pain levels using EPIC questionnaire | 2 years
  Pain levels will be collected using expanded prostate cancer index composite (EPIC) questionnaire. The quality-of-life scores will be converted to a scale of 0-100 for each category. A higher score indicates a better quality of life.
Urinary function using EPIC questionnaire | 2 years
  Urinary function will be collected using expanded prostate cancer index composite (EPIC) questionnaire. The quality-of-life scores will be converted to a scale of 0-100 for each category. A higher score indicates a better quality of life.
Bowel function using EPIC questionnaire | 2 years
  Bowel function will be collected using expanded prostate cancer index composite (EPIC) questionnaire. The quality-of-life scores will be converted to a scale of 0-100 for each category. A higher score indicates a better quality of life.
Assessment of adaptive RT approach using dose accumulation | 2 years
  Dosimetric assessment of the CBCT-guided online adaptive RT approach using dose accumulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada